CLINICAL TRIAL: NCT00089414
Title: The Treatment of Menstrually-Related Mood Disorders With Extended Versus Interrupted Oral Contraceptives
Brief Title: Treatment of Menstrually Related Disorders With Continuous v. Interrupted Oral Contraceptives
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Informed by manufacturer that CDB-2914 crosses blood-brain barrier invalidating Arm #3 of protocol.
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 040221; 04-M-0221
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Results first posted 2017-01-02 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-07

CONDITIONS: Premenstrual Syndrome; PMS; Premenstrual Dysphoric Disorder; PMDD; Depression
Keywords: Depression; Menstrual Cycle; Gonadal Steroids; Ethinyl Estradiol; Drospirenone; Menstrually Related Mood Disorder; MRMD
MeSH Terms: conditions — Premenstrual Syndrome; Premenstrual Dysphoric Disorder; Depression | interventions — drospirenone and ethinyl estradiol combination; ulipristal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Treatment arm # 1 consists of the continuous administration of Yasmin oral contraceptive (a combination of 30 µg of ethinyl estradiol and 3 mg of drospirenone) for 15 weeks starting on day 2 to 5 of the first menstrual cycle.
  Interventions: Drug: Ethinyl Estradiol/Drospirenone
- 2 (Active Comparator): Treatment arm # 2 (interrupted Yasmin administration) will be identical to arm # 1 with the exception that the continuous administration of Yasmin will be interrupted by the substitution of placebo for Yasmin for one week during weeks 3, 8, and 14 of the study. The women participating in this treatment arm will experience episodes of menstruation after Yasmin withdrawal (when they are on placebo).
  Interventions: Drug: Ethinyl Estradiol/Drospirenone; Drug: Placebo
- 3 (Active Comparator): Yasmin oral contraceptive; CDB 2914 progesterone antagonist. Treatment arm # 3 is identical to treatment arm # 1 with the exception that the continuous administration of Yasmin will also include the administration of progesterone antagonist CDB-2914 during weeks 3, 8, and 14. Menses is anticipated to occur within 2-3 days of CDB-2914 administration. Women in treatment arms # 3 and # 1 will be exposed to continuous levels of Yasmin, but due to the local effects of the progesterone antagonist on the endometrium, women in arm # 3 will experience menses.
  Interventions: Drug: Ethinyl Estradiol/Drospirenone; Drug: CDB 2914

INTERVENTIONS:
Drug: Ethinyl Estradiol/Drospirenone — Drug administered dependent upon arm.
  Other Names: Yasmin
Drug: Placebo
  Arms: 2
Drug: CDB 2914
  Other Names: Progesterone antagonist
  Arms: 3

SUMMARY:
This study will determine whether uninterrupted treatment with birth control pills over several menstrual cycles prevents severe premenstrual syndrome (PMDD).

Previous studies have shown that the hormones estrogen and progesterone regulate mood in women with MRMD. This study will use various treatment regimens with birth control pills and placebo (sugar pill) to clarify the relationships among estrogen and progesterone, the menstrual cycle, and mood.

Healthy women between 18 and 45 years of age who menstruate may be eligible for this 15-week study. Candidates are screened with a physical examination, blood and urine tests, an electrocardiogram, and 3 months of symptoms ratings to confirm MRMD.

Participants are randomly assigned to one of three treatment groups. Group 1 takes a birth control pill every day and on three occasions takes a placebo capsule. Group 2 takes a birth control pill most but not all days and on three occasions takes a placebo capsule. Group 3 takes a birth control pill every day and on three occasions takes another medication called CDB-2914 that causes menstrual bleeding to occur.

Participants come to the NIH clinic every other week for blood tests and measurement of vital signs (blood pressure, pulse, and temperature) and to complete symptoms ratings scales. Subjects who develop breakthrough bleeding (menstruation earlier than expected) will have a transvaginal ultrasound. For this procedure, a probe is inserted into the vagina for about 10 minutes. The probe gives off and receives sound waves that can be used to form a picture of the endometrium (lining of the uterus).

...

DETAILED DESCRIPTION:
Results from previous protocols (#90-M-0088 and 92-M-0174) have demonstrated that women with menstrually-related mood disorder (MRMD), but not women lacking this disorder, experience mood deterioration within approximately one to two weeks after exposure to either estradiol or progesterone in the context of gonadal suppression (induced by use of the depot gonadotropin releasing hormone agonist leuprolide acetate). Preliminary results of protocol 00-M-0103 suggest that this hormone-induced depression occurs consequent to changes in gonadal steroid levels and not to simple exposure to basal levels above a critical threshold. Additionally, continued administration of hormone for three months resulted in no further symptoms subsequent to the initial precipitated episode. These data suggest the potential therapeutic benefit of extended oral contraceptive (OC) regimens with reduced pill-free intervals in MRMD to minimize the mood destabilizing effects of changing hormone levels. In this protocol we examine whether the effects of 15 weeks of continuous oral contraceptive administration causes a remission of symptoms in women with MRMD.

ELIGIBILITY:
* INCLUSION CRITERIA (are from protocol 81-M-0126 and are as follows):
* Subjects who meet criteria for MRMD are healthy (by physical exam, normal pelvic exam and pap smear, and normal lab values) and medication free will be included in this study.
* Oral contraceptives (and CDB-2914 in arm #3) will not be administered to any subject with significant clinical or laboratory abnormalities.

EXCLUSION CRITERIA:

Any patient with a current axis I psychiatric diagnosis will be excluded from participating in this protocol.

Subjects taking psychotropic agents (e.g. antidepressants, anxiolytics or mood stabilizers) will likewise be excluded from the study.

Women who have received glucocorticoid or megestrol therapy within the last year (and thus may experience residual suppression of the compensatory HPA axis response to CDB-2914-induced glucocorticoid receptor antagonism) will be also excluded, albeit almost entirely on theoretical grounds.

Women who have any chronic medical conditions or are taking medications will be excluded.

Women who have a medical condition or are taking any chronic medications that may increase serum potassium levels will also be excluded.

Those patients who would be uncomfortable with extending the length of their menstrual cycles will not be enrolled in this study and will either be offered participation in another study or an outside referral for treatment in the community.

The following conditions will constitute contraindications to treatment with continuous oral contraception or the use of the progesterone antagonist, CDB-2914, and will preclude a patient's participating in this protocol:

* history of endometriosis, or recent, rapid growth of uterine fibroid tumors (defined as doubling in size in six month period);
* diagnosis of ill-defined, obscure pelvic lesions, particularly undiagnosed ovarian enlargement;
* hepatic disease as manifested by abnormal liver function tests;
* history of breast carcinoma;
* history of pulmonary embolism or phlebothrombosis;
* undiagnosed vaginal bleeding;
* porphyria;
* history of malignant melanoma;
* history of cholecystitis or pancreatitis;
* history of hypercholesterolemia, hypertension, diabetes, or renal disease;
* recurrent migraine headaches (greater than or equal to 3 per year) in women 35 or older;
* pregnancy or lactation;
* cigarette smoking in women 35 or older, or more than 10 cigarettes per day in women under 35; or
* use of oral, injectable, or inhaled glucocorticoids or megestrol within the last year.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2004-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro E Martinez, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Backstrom T, Sanders D, Leask R, Davidson D, Warner P, Bancroft J. Mood, sexuality, hormones, and the menstrual cycle. II. Hormone levels and their relationship to the premenstrual syndrome. Psychosom Med. 1983 Dec;45(6):503-7. doi: 10.1097/00006842-198312000-00004. PMID 6686333
- [Background] Schmidt PJ, Nieman LK, Grover GN, Muller KL, Merriam GR, Rubinow DR. Lack of effect of induced menses on symptoms in women with premenstrual syndrome. N Engl J Med. 1991 Apr 25;324(17):1174-9. doi: 10.1056/NEJM199104253241705. PMID 2011161
- [Background] Muse KN, Cetel NS, Futterman LA, Yen SC. The premenstrual syndrome. Effects of "medical ovariectomy". N Engl J Med. 1984 Nov 22;311(21):1345-9. doi: 10.1056/NEJM198411223112104. PMID 6387488

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Yasmin: Treatment arm # 1 consists of the continuous administration of Yasmin oral contraceptive (a combination of 30 µg of ethinyl estradiol and 3 mg of drospirenone) for 15 weeks starting on day 2 to 5 of the first menstrual cycle.
- Interrupted Yasmin: Treatment arm # 2 (interrupted Yasmin administration) will be identical to arm # 1 with the exception that the continuous administration of Yasmin will be interrupted by the substitution of placebo for Yasmin for one week during weeks 3, 8, and 14 of the study. The women participating in this treatment arm will experience episodes of menstruation after Yasmin withdrawal (when they are on placebo).
- Continuous Yasmin Plus Progesterone Antagonist: Yasmin oral contraceptive; CDB 2914 progesterone antagonist. Treatment arm # 3 is identical to treatment arm # 1 with the exception that the continuous administration of Yasmin will also include the administration of progesterone antagonist CDB-2914 during weeks 3, 8, and 14. Menses is anticipated to occur within 2-3 days of CDB-2914 administration. Women in treatment arms # 3 and # 1 will be exposed to continuous levels of Yasmin, but due to the local effects of the progesterone antagonist on the endometrium, women in arm # 3 will experience menses.
Period: Overall Study
Arm/Group | Continuous Yasmin | Interrupted Yasmin | Continuous Yasmin Plus Progesterone Antagonist
Started | 2 | 1 | 2
Completed | 2 | 1 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Continuous OCP Plus Placebo: Treatment arm # 1 (extended ethinyl estradiol and progestin [EE/P]) consists of the continuous administration of 30 µg of ethinyl estradiol and 3 mg of drospirenone (Yasmin) for 15 weeks starting on day 2 to 5 of the first menstrual cycle.
- Interrupted OC: Treatment arm # 2 (interrupted EE/P administration) will be identical to arm # 1 with the exception that the continuous administration of EE/P will be interrupted by the substitution of placebo for EE/P for one week during weeks 3, 8, and 14 of the study. The women participating in this treatment arm will experience episodes of menstruation after EE/P withdrawal (placebo).
- Continuous OC Plus PR Antagonist: Yasmin oral contraceptive; CDB 2914 progesterone antagonist. Treatment arm # 3 (extended EE/P with menses) is identical to treatment arm # 1 except the progesterone antagonist CDB-2914 will be administered during weeks 3, 8, and 14. Menses is anticipated to occur within 2-3 days of CDB-2914 administration. As such, menses will occur in these women at approximately the same interval as experienced by those women in treatment arm # 2 due to the local effects of the progesterone receptor antagonist on the endometrium (lining of the uterus). Thus, women in treatment arms # 3 and # 1 will be exposed to continuous levels of ethinyl estradiol and progestin, but due to the local effects of the progesterone antagonist on the endometrium, women in arm # 3 will experience menses.
- Total: Total of all reporting groups
Arm/Group | Continuous OCP Plus Placebo | Interrupted OC | Continuous OC Plus PR Antagonist | Total
Number analyzed (Participants) | 2 | 1 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 2 | 5
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (6.364) | 41 (0) | 34.5 (2.121) | 34.6 (3.8794)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 5
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 2 | 5

OUTCOME MEASURES:

1. Secondary Outcome: Change in Clinical Global Impression Scale (CGI) Factors Associated With Premenstrual Symptoms.
Description: The CGI was developed for use in NIMH-sponsored clinical trials to provide a brief, stand-alone assessment of the clinician's view of the patient's global functioning prior to and after initiating a study medication.1 The CGI provides an overall clinician-determined summary measure that takes into account all available information, including a knowledge of the patient's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the patient's ability to function. The CGI actually comprises two companion one-item measures evaluating the following: (a) severity of psychopathology from 1 to 7 and (b) change from the initiation of treatment on a similar seven-point scale, with 1 being normal/more improved and 7 being severe/worse.
Time Frame: Every 2 wks for 3 months
Population: This study was terminated early due to confounding factors in design. Protocol terminated after receiving information from manufacturer (Pharma) that CDB-2914 crosses the blood-brain barrier, invalidating Arm #3 due to potential Central Nervous System effect of the compound on behavior.
Arm/Group | Continuous Yasmin | Interrupted Yasmin | Continuous Yasmin Plus Progesterone Antagonist
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Change in Premenstrual Tension Syndrome Scale (PMTS) Factors Associated With Premenstrual Symptoms.
Description: The PMTS observer scales assess symptoms in ten different domains including irritability-hostility; tension; efficiency; dysphoria; moodiness; motor coordination; mental-cognitive functioning; eating habits; sexual drive and activity; physical symptoms and social impairment. They have been used to measure premenstrual symptom severity and response to treatment in several clinical trials and prevalence studies. Score ranges from no symptoms to severe symptoms on a scale of 0 to 6, with 0 being no symptoms and 6 being severely symptomatic.
Time Frame: Every 2 weeks for 3 months
Population: as for outcome 1
Arm/Group | Continuous Yasmin | Interrupted Yasmin | Continuous Yasmin Plus Progesterone Antagonist
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change in Beck Depression Inventory (BDI) Factors Associated With Premenstrual Symptoms
Description: The Beck Depression Inventory (BDI)is a 21-question multiple-choice self-report inventory, one of the most widely used instruments for measuring the severity of depression. Total scores are interpreted per these ranges:
  0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression.
Time Frame: Every 2 weeks for 3 months
Population: as for outcome 1
Arm/Group | Continuous Yasmin | Interrupted Yasmin | Continuous Yasmin Plus Progesterone Antagonist
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Continuous OCP Plus Placebo | Interrupted OC | Continuous OC Plus PR Antagonist
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/2

LIMITATIONS AND CAVEATS:
Protocol terminated after receiving information from manufacturer (Pharma) that CDB-2914 crosses the blood-brain barrier, invalidating Arm #3 due to potential CNS effect of the compound on behavior.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes